CLINICAL TRIAL: NCT02051192
Title: A Brief Behavioral Treatment for Anxiety in Young Children
Brief Title: Brief Behavioral Treatment for Anxiety in Young Children
Acronym: PLET
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Adam Lewin, Assistant Professor, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PLET-13-0634
Record Dates: First submitted 2014-01-29; First posted 2014-01-31 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-10

CONDITIONS: Obsessive-compulsive Disorder; Social Phobia; Generalized Anxiety Disorder; Specific Phobia; Separation Anxiety Disorder; Selective Mutism; Anxiety Disorder, Not Otherwise Specified
Keywords: obsessive-compulsive disorder; Social phobia; Generalized anxiety disorder; Specific phobia; Separation anxiety disorder; Selective Mutism; Anxiety Disorder, Not Otherwise Specified; Counseling; Behavioral therapy; Psychotherapy; Exposure; Young Children
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Phobia, Social; Generalized Anxiety Disorder; Phobia, Specific; Anxiety, Separation; Mutism; Anxiety Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Parent-Led Exposure Therapy (PLET) (Experimental): Therapists will work with families for 10 sessions, twice weekly. The first treatment session will be a 90 minute parent only psychoeducation and treatment preparation session. Each subsequent session will last up to 60 minutes and will consist of exposure therapy using developmentally appropriate modulated behavioral approaches such as Participant modeling (PM) and Reinforced practice (RP).
  Interventions: Behavioral: Parent-Led Exposure Therapy
- Treatment As Usual (Active Comparator): Patients randomized to the TAU arm will be instructed to continue receiving their prior interventions as recommended by their providers (e.g., psychotherapy, social skills training, behavioral interventions, family participation in family therapy or a parenting class, or pharmacological interventions). Treatment changes (e.g., medication increase, starting psychotherapy in the community) are not prohibited and will be monitored. Thus, treatment will continue as it would in standard practice.
  Interventions: Other: Treatment As Usual

INTERVENTIONS:
Behavioral: Parent-Led Exposure Therapy — Therapists will work with families for 10 sessions, twice weekly. The first treatment session will be a 90 minute parent only psychoeducation and treatment preparation session. Each subsequent session will last up to 60 minutes and will consist of exposure therapy using developmentally appropriate modulated behavioral approaches such as Participant modeling (PM) and Reinforced practice (RP).
  Other Names: Brief Behavioral Treatment for Anxiety in Young Children
  Arms: Parent-Led Exposure Therapy (PLET)
Other: Treatment As Usual — Patients randomized to the TAU arm will be instructed to continue receiving their prior interventions as recommended by their providers (e.g., psychotherapy, social skills training, behavioral interventions, family participation in family therapy or a parenting class, or pharmacological interventions). Treatment changes (e.g., medication increase, starting psychotherapy in the community) are not prohibited and will be monitored. Thus, treatment will continue as it would in standard practice. These participants may also elect to receive no treatment at all during the TAU period.
  Arms: Treatment As Usual

SUMMARY:
Behaviorally and cognitive-behaviorally based therapeutic techniques (BT; CBT) that incorporate exposure therapy useful for treatment of anxiety disorders among typically developing children. Although a large amount of data demonstrate the effectiveness of of BT and CBT approaches for treating anxious youth, there is a gap in the literature for the effectiveness of these approaches for children under the age of seven. Evidence increasingly suggests that family factors such as accommodation and parenting style contribute significantly to the presence of anxiety symptoms as well as treatment outcomes, particularly in young children. These findings stress the importance of using a treatment approach in which parents are directly involved in education, parent training, and generalization of treatment effects. Therefore, this study aims to evaluate a new treatment program, parent-led behavioral treatment, for children ages 3 to 7 years of age who have a principal anxiety disorder diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient children between the ages 3-7 years.
* Meets DSM-IV criteria for a primary diagnosis of an anxiety disorder or achieves a minimum score of 12 Pediatric Anxiety Rating Scale (PARS)
* Child has a PPVT IV SS > 80.
* Patients with co-morbid depression, ADHD, tic disorder or disruptive behavior disorders will be included as long as anxiety is primary (i.e., most impairing/distressing).

Exclusion Criteria:

* • (a) Current clinically significant suicidality or (b) individuals who have engaged in suicidal behaviors within 6 months will be excluded and referred for appropriate clinical intervention.

  * Receiving concurrent psychotherapy, social skills training, or behavioral interventions (e.g., applied behavior analysis). Families will have the option of discontinuing such services to enroll in the study. Those randomized treatment as usual (TAU) will be able to continue or initiate psychosocial interventions (psychotherapy, social skills training, applied behavior analysis, or family therapy) whereas those randomized to PLET will not receive these interventions concurrent with PLET.
  * Any change in established psychotropic medication (e.g., antidepressants, anxioloytics, antipsychotics, stimulants) within 10 weeks before study. Those randomized to TAU may make medication changes following randomization, including starting a medication; those randomized to PLET will remain stable on medications during the study.
  * Absence of language.
  * A formal diagnosis of mental retardation or autism spectrum disorder.
  * Unwillingness of parents to make the commitment to accompany their child for multiple study visits, unwillingness to take part in randomization, inability to attend sessions twice weekly as therapist availability allows, inability to attend assessment visits.
  * Presence of a significant and/or unstable medical illness which might lead to hospitalization during the study.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2014-01; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Pediatric Anxiety Rating Scale | after 5 weeks of treatment
  The PARS is a clinician-rated scale assessing anxiety symptoms and the associated severity and impairment in children over the past week.
Clinical Global Impression - Severity | After 5 weeks of treatment
  The CGI-S is a 7-point clinician rating of severity of psychopathology anchored by 1 ("no illness") and 7 ("very severe").
Clinical Global Improvement | After 5 weeks of treatment
  The CGI is a 7-point rating of treatment response anchored by 1 ("very much improved) and 7 ("very much worse"). Youth being rated by the IE as 1 ("very much improved") and 2 ("much improved") will be considered treatment responders.

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Center for Pediatric Neuropsychiatry - University of South Florida, St. Petersburg, Florida, United States